CLINICAL TRIAL: NCT07216300
Title: OMT for Overhead Throwing Performance: A Study on Shoulder and Hip Interventions
Brief Title: Osteopathic Manipulative Treatment for Pitch Performance in Baseball Players: A Study on Shoulder and Hip Interventions
Acronym: PITCH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: William Carey University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB #2025-067
Record Dates: First submitted 2025-10-02; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pitch; Baseball Pitcher; Throwing Performance
Keywords: osteopathic; pitcher; pitch performance; baseball; college sports
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: This study will be a randomized control trial. If there is insufficient statistical power, then the control subjects will be rolled into the intervention arm of the study at 5 weeks (+/-2 depending on the calendar), and the study will convert to a prospective cohort design. RCT was chosen because it is the gold standard for researching a medical intervention. The back-up plan is necessary because the maximum available cohort is limited by the size of the William Carey baseball team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control grop (No Intervention): no intervention, solely measurement of pitch metrics and arm ranges of motion
- experimental (Experimental): OMT intervention, and measurement of pitch metrics and arm ranges of motion
  Interventions: Procedure: Osteopathic Manipulative Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Manual Medicine applied either by a physician or a medical student
  Arms: experimental

SUMMARY:
To investigate the impact of manual medicine on key aspects of the kinetic chain on measures of performance in baseball players.

DETAILED DESCRIPTION:
An OMT protocol which targets the hips, diaphragm, and throwing shoulder will be investigated for improvement to pitch metrics of the fastball in the experimental group compared with the control group. OMT protocol is expected to increase the active ranges of motion of the throwing shoulder and the bilateral hips of those in the experimental group compared to the control group. Kerlan-Jobe Orthopaedic Clinic Shoulder and Elbow Score (KJOC-SES) will also improve in the experimental group compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Presently on the William Carey University baseball team
* Permission granted by the coach for participation
* Sports physical completed clearing the subject for participation in sports for the academic year

Exclusion Criteria:

* injuries which prevent the subject from participation in practice and in games

Ages: 18 Years to 102 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-14 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Pitch Metrics: Speed | 5 weeks
  Velocity in miles per hour, Effective Velocity in miles per hour
Shoulder and Hip Ranges of Motion | 5 weeks
  GH Internal Rotation in degrees, GH External Rotation in degrees, GH Flexion in degrees, GH Extension in degrees, GH abduction in degrees, Hip flexion in degrees, Hip Extension in degrees, Hip Internal Rotation in degrees
Pitch Metrics: Spin | 5 weeks
  Ball spin in revolutions per minute
Pitch Metrics: Zone time | 5 weeks
  Zone time in seconds
Pitch Metrics: Ball movement | 5 weeks
  Horizontal Break in inches, Vertical Break in inches, Induced Vertical break in inches
Pitch Metrics: Pitcher Mechanics | 5 weeks
  Pitch Extension in inches

SECONDARY OUTCOMES:
Kerlan-Jobe Orthopaedic Clinic (KJOC) Shoulder and Elbow Score Calculator | 5 weeks
  Shoulder Elbow Score, subjective measure of performance, measured in points (per the survey) with higher values corresponding to improved function and lower values reflecting limited function

CONTACTS AND LOCATIONS:
Locations (1):
- William CArey University, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol, and deidentified individual raw data
Supporting Information: Study Protocol
Time Frame: Available beginning Oct 2025 and continuing for 4 years
Access Criteria: Contact Carissa Rosten of Danielle Fastring and request deidentified information on excel sheets, and protocol can be shared within the IRB submission packket